CLINICAL TRIAL: NCT01160068
Title: A Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Bioequivalence Study of Metformin Hydrochloride 1000 mg Tablets (Dr. Reddy's Laboratories Ltd., Generics, India) to be Compared With Glucophage® (Metformin Hydrochloride) 1000 mg Tablets (Bristol-Myers Squibb, USA) in 48 + (2 Standby) Healthy, Adult, Human Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Metformin Hydrochloride Tablets 1000 mg Tablets of Dr. Reddy's Laboratories Limited Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Vice President-Generics, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8322
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2005-01

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin Hydrochloride 1000 mg tablets of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Metformin
- Glucophage (Active Comparator): Glucophage 1000 mg tablets of Bristol-Myers Squibb
  Interventions: Drug: Glucophage

INTERVENTIONS:
Drug: Metformin — Metformin Tablets 1000 mg
  Other Names: Glucophage Tablets 1000 mg
  Arms: Metformin
Drug: Glucophage — Glucophage 1000 mg tablets of Bristol-Myers Squibb
  Arms: Glucophage

SUMMARY:
To compare the single dose bioavailability of Metformin Hydrochloride 1000 mg tablets (Dr. Reddy's Laboratories Ltd., Generics, India) with Glucophage (Metformin Hydrochloride) 1000 mg tablets (Bristol-Myers Squibb, USA) in 48 + (2 standby) healthy, adult, human subjects under fed conditions.

To monitor adverse events and to ensure the safety of subjects.

DETAILED DESCRIPTION:
Open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose,crossover bioequivalence study with at least 07 days of washout period between each drug administration under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provided written informed consent.
* Subjects who were healthy within 18-45 years of age (inclusive) weighing at least 50 kg.
* Subjects who were within ±10% of ideal body weight in relation to height according to Life Insurance Corporation of India height-weight chart for non-medical cases.
* Subjects with normal health as determined by medical history and physical examination performed within 15 days prior to the commencement of the study.
* Subjects with normal ECG, X-ray and vital signs.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent
* If subject is a female volunteer and

  * is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device(IUD), or abstinence.
  * is postmenopausal for at least 1 year.
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

* Subjects incapable of understanding the informed consent.
* Subjects with BP:≤90/60 or BP≥140/90.
* History of hypersensitivity or idiosyncratic reaction to Metformin or other Biguanides.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal, endocrine, immunologic, neurologic and haematologic function.
* Regular smoker who smokes more than ten cigarettes daily and has difficulty in abstaining from smoking for the duration of each study period.
* Subjects who has taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication within the past 30 days prior to start of clinical period.
* History of any psychiatric illness, which may impair the ability to provide written, informed consent.
* Subjects who have a history of alcohol or substance abuse within the last 5 years.
* Subjects with clinically significant abnormal values of laboratory parameters.
* Subjects who have participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
* Subjects who tested positive at screening for HIV, HbsAg or HCV
* Subjects with positive urine drug screen test for drugs of abuse.
* Any subject in whom Metformin is contraindicated for medical reasons.
* Subjects who have used any drugs or substances such as herbal preparations known to be strong inhibitors of CYP enzymes (formerly known as cytochrome P450 enzymes) within 14 days prior to the first dose.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breast-feeding.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax, AUC, Tmax,t1/2 parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mangesh Kulkarni, MD, Principal Investigator — Vimta Labs Ltd.
Locations (1):
- Vimta Labs Ltd., Hyderabad, Andhra Pradesh, India